CLINICAL TRIAL: NCT04376372
Title: Forced Lefthandedness in Neonatal Brachial Plexus Palsy (NBPP) Children : is There a Neurophysiological and Functional Difference With Natural Lefthanders
Brief Title: Forced Lefthandedness in Neonatal Brachial Plexus Palsy (NBPP) Children
Acronym: NBPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201525721
Record Dates: First submitted 2020-04-15; First posted 2020-05-06 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Neonatal Brachial Plexus Palsy
Keywords: upper limb paresis; developmental; functiona laterality
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy; Paresis | interventions — Magnetic Resonance Imaging; Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TD_lefthanders: Typical developing lefthanded children and adolescents Assessment : sensibility, strength,writing,manual dexterity,degree of lefthandedness, body representation, movement analysis, motor control, quality of life, participation
  Interventions: Diagnostic Test: Functional testing, Magnetic resonance imaging, Electromyography
- F_lefthanders: Forced left handed NBPP children Assessment : sensibility, strength,writing,manual dexterity,degree of lefthandedness, body representation, movement analysis, motor control, quality of life, participation
  Interventions: Diagnostic Test: Functional testing, Magnetic resonance imaging, Electromyography

INTERVENTIONS:
Diagnostic Test: Functional testing, Magnetic resonance imaging, Electromyography — Electromyography only for cases (F-Lefthanders), not for controls (TD-lefthanders)

SUMMARY:
The aim of the project is to assess the neurophysiological and functional consequences of forced lefthandedness in a population with right neonatal brachial plexus palsy (NBPP).

DETAILED DESCRIPTION:
A cross-sectional case-control study design to assess the neurophysiological and functional consequences of forced lefthandedness in a population with right neonatal brachial plexus palsy (NBPP). Controls are natural lefthanded typical developing children and adolescents.Case and controls are matched for age, gender and activity level.

ELIGIBILITY:
Inclusion Criteria:

* typical developing
* lefthanded
* NBPP or healthy
* righthanded parents
* 6-23 years

Exclusion Criteria:

* history of other locomotor or neurological disorder than NBPP
* history of brain surgery
* history of psychiatric disorder

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Group 1 : healthy lefthanded typical developing children and adolescents with righthanded parents Group 2 : Forced lefthanded NBPP children and adolescents with righthanded parents
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Strength-1 | Baseline
  Medical Research Council Scale (MRC-scale) : score 0-5 ; 0 : no muscle contraction (worse) to 5 : normal power (better)
Strength-2 | Baseline
  Grip Strength (E-link) : Percent of the norm : higher = better
Strength-3 | Baseline
  Active Movement scale (AMS): score 0-7 ; 0: no contraction to 7 : full motion
Sensibility hand | Baseline
  Semmes-Weinstein monofilament ( normal- abnormal)
Handedness | Baseline
  Edinburgh Handedness Inventory (EDI) : Lateralization index: -100 (pure lefthander) to +100 (pure righthander)
Baseline measure : brain imaging | Baseline
  Magnetic resonance imaging (MRI)
Baseline measure : movement pattern | Baseline
  Kinematic movement analysis (kinematic angels, kinetic forces, movement patterns)
Body representation | Baseline
  actual, implicit hand representation by drawings : mm

SECONDARY OUTCOMES:
quality of life-1 | Baseline
  the Pediatric Outcome Data Collecting Instrument - dutch version
  • The PODCI consists of 5 domains: Upper Extremity and Physical Function, Transfers and Basic Mobility, Sports and Physical Functioning, Pain/Comfort, and Happiness. The "Global Functioning Score" is a mean of all domains except Happiness. The PODCI divides the ages into 2 groups: ages 2 to 10 years, which is filled out by the parent/guardian only, and ages 11 to 18 years, which has a questionnaire to be filled out by both the parents/guardians and the child. A raw score is created both for each domain and for the Global score, and can be compared with a normative standard
quality of life-2 | Baseline
  KIDSCREEN-52- dutch version : questionnaire of 52 items to be answered by the child/adolescent assessing Health related Quality of Life. • The KIDSCREEN items use 5-point Likert-type scale. Rasch scores are computed for each dimension and transformed into T-values with a mean of 50 and a standard deviation of 10; higher scores indicate better HRQoL and well-being.KIDSCREEN-52 T scores refer to the mean values and standard deviations from a multinational European sample
Activity-1 | Baseline
  The Children's Hand-use Experience Questionnaire (CHEQ) is an online questionnaire for children from 6 to 18 years with unilateral upper limb impairment. It is designed to measure children's own experiences when using the affected hand in common daily life activities requiring use of both hands.For children below the age of 13 years, it is recommended that parents act as proxy. CHEQ is a computer-adaptive online questionnaire consisting of 29 items; available free of charge via the website (www.cheq.se). Three scales are used to measure the grasp efficacy when both hands are involved, time utilization when performing the activity compared with peers, and experience of feeling bothered while performing the activities independently. CHEQ scales are rated on a four-point ordinal scale and raw scores can be transformed by Rasch analysis to logits and further into a 0-100 CHEQ-units;Higher scores indicate a better grasp, less time taken, and greater satisfaction.
Activity-2 | Baseline
  Assisting Hand assessments (AHA). The AHA is used to score object-related hand actions observed during a semi-structured test situation (10-20min) that elicits the use of both hands and which is suitable for different age groups.A transformation table of raw scores to interval-level 'AHA units' is available. (0-100). The higher the score the more the hand is properly used as assisted hand
Activity-3 | Baseline
  The Melbourne Assessment is based on 16 items comprising tasks that are representative of the most important components of unilateral upper limb function (reach, grasp, release, and manipulate). Most items are further subdivided in two to four sub-items that represent an aspect of the required movement, such as range of movement, fluency, target accuracy, speed, and quality of movement. The total score can range from 0 to 122 points and can be converted to a percentage. The higher the score, the better the unilateral limb function
Activity-4 | Baseline
  The Purdue Pegboard Test is designed to assess fine motor hand function. This assessment involves a series of four subtests that consist of placing small pins into holes on a pegboard and assembling pins and washers. The subsets for preferred, non-preferred, and both hands require the patient to place the pins in the holes as quickly as possible, with the score being the number of pins placed in 30 s. Aged normed data are available.
shoulder function cases | Baseline
  mallet scale of shoulder function : 8 items. In the Mallet score, shoulder movements are graded on a scale from 1 (no motion) to 5 (normal motion equal to that in the unaffected side), resulting in a maximum total score of 40. A Mallet subscore of 4 or better is considered to be good shoulder function
Function( for cases) | Baseline
  Brachial plexus outcome measure (BPOM) :The BPOM is a, disease-specific, functional upper extremity assessment for children with NBPP. It has 2 subscales: Activity and Self-evaluation. The BPOM Activity subscale has 11 items, and each item is scored between 1 and 5 on an ordinal scale. A score of1 indicates that the task cannot be completed, and a score of 5 indicates that the task can be completed with normal movement pattern. The Activity subscale contains 3 parts: (1) shoulder, (2) elbow and forearm, and (3) wrist, finger, and thumb. The BPOM Self-evaluation subscale consists of 2 visual analog scales to evaluate the working of the arm and hand and 1 visual analog scale to evaluate the appearance of the arm and hand of the child. Several categories and items are evaluated simultaneously, and each score is calculated separately to define the function
cognition | baseline
  Wechsler intelligence Scale for children: a short form consisting of subtests : (picture completion (PC), Vocabulary (V), Block Design (BD) and Similarities (S))of the WISC-III to estimate participant's intelligence.
  The subtest scores of the short form were transformed into deviation IQs (DIQ), based on mean intercorrelations from the standardization sample (Wechsler, 1991).
  • Classification : volgens DIQ
  * < of = 89 : below average
  * 90 of = 109 : average
  * 110 of > : above average
muscle and nerve function | baseline
  electromyography (EMG)
writing | baseline
  Vlaamse schrijftest : norms per age

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Van der Looven, MD, Principal Investigator — Physical Medicine and Rehabilitation
Locations (1):
- Physical Medicine and Rehabilitation, Ghent, Oost Vlaanderen, Belgium